CLINICAL TRIAL: NCT01909726
Title: The Art of Waiting: Evaluation of an Interactive Media Experience in a Children's Hospital Clinic Waiting Space
Status: Completed | Type: Observational
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: BloorviewKR
Record Dates: First submitted 2013-01-30; First posted 2013-07-26 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2014-07

CONDITIONS: Anxiety
Keywords: Hospital Design; Technology; Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Interactive media: ScreenPlay
  Interventions: Other: ScreenPlay
- Passive media: Silent nature video
- No media: Standard care

INTERVENTIONS:
Other: ScreenPlay — Interactive technology
  Groups: Interactive media

SUMMARY:
The purpose of this study is to test the hypothesis that providing low-intensity opportunities for interactive play can improve the waiting and overall clinic experiences of children. This study evaluates an innovative, interactive system called ScreenPlay designed to realize the intentions of the "Healing Environment" in the waiting space of a paediatric hospital.

DETAILED DESCRIPTION:
Existing entertainment and distraction options (e.g. toys, video games) meet neither organizational standards nor families' needs with respect to accessibility and infection control. Additionally, they do not provide the types of positive experiences (e.g. calm, low intensity) that are most desirable for children awaiting treatment.

The goal of this research is to empirically evaluate the effectiveness of ScreenPlay, a technology that enables users to create or manipulate animations on a screen/projection, and to provide an evidence-informed model for the design of optimal paediatric waiting spaces. A blinded, clustered, parallel randomized controlled trial applying objective outcome measures and qualitative methods will be used to compare children allocated to one of three waiting conditions at a large urban rehabilitation hospital: (a) no media (standard care), (b) passive media (a silent nature video), or (c) interactive media (ScreenPlay). This study will answer the questions:

Can Interactive Media (i.e. ScreenPlay):

1. reduce state anxiety in children/youth attending an outpatient clinic? and,
2. improve child, parent, and staff satisfaction with the clinic experience?

We hypothesize that:

1. Decreases in state anxiety will be greater for children exposed to ScreenPlay for 10 minutes than for those exposed to passive (i.e. a nature video) or no media (i.e. standard care/control). The decrease in state anxiety associated with ScreenPlay will be >5 points on the normalized 100 point State Anxiety Scale.
2. ScreenPlay will generate more movement/activity on the floor (i.e. an indicator of active engagement with the system) than the passive media or control conditions as measured via contact floor sensors.
3. The waiting and overall clinic experience of children with diverse mobility, parents, and staff will be perceived more positively when exposed to ScreenPlay as compared to passive media or control conditions.

ELIGIBILITY:
Participants include clients, their parents/guardians, and staff associated with the outpatient clinic at Holland Bloorview Kids Rehabilitation Hospital.

1. Children and youth aged 5 to 19 years and their guardian/parent.
2. Anticipated wait time ≥30 minutes to allow time to complete the study.
3. Ability to communicate in English through speech, writing/typing, or other communication device. Note: For children who cannot communicate their thoughts/feelings, parent-proxy may be used.
4. All outpatient clinic staff

Ages: 5 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants include clients, their parents/guardians, and staff associated with the outpatient clinic at Holland Bloorview Kids Rehabilitation Hospital.
Sampling Method: Probability Sample
Enrollment: 310 (Actual)
Dates: Start 2012-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
State Trait Anxiety Inventory, STAI | Baseline, after 10 minutes of exposure to intervention, and immediately following appointment.
  The STAI is used to capture apprehension, tension, nervousness, and worry.

SECONDARY OUTCOMES:
Modified Yale Preoperative Anxiety Scale, mYPAS | Baseline, after 10 minutes of exposure to intervention, and immediately following appointment.
  The mYPAS observes activity, vocalizations, emotion expressivity, state of arousal, and use of parents, to ascertain children's anxiety state.
Faces Pain Scale Revised, Faces-R | Immediately following medical/therapeutic intervention.
  Faces-R is used to capture self-reported pain. The scale is composed of 6 gender neutral faces showing increasing levels pain/hurt from "no pain" to "most pain possible"

OTHER OUTCOMES:
Behaviour Mapping | Administered during the participant's 10 minute exposure to the intervention.
  An unobtrusive, observational technique used to systematically define/record distinct behaviours including: mobility, activities, social interactions, emotion expressivity, attention/engagement, and description of challenges encountered.
Contact sensors | Data from sensors is continuously collected from 7am to 5pm from beginning of data collection (June 2012) to end of data collection (April 2013)
  ScreenPlay incorporates a 'pressure' floor composed of 100 contact sensors arranged in a 10 foot by 10 foot grid. Activity metrics (e.g. number, duration, and frequency of activations) are extracted for each contact sensor and for the amalgamated grid.
Feedback questionnaires | Child and parent surveys are administered post-exposure. Staff surveys will be administered nearing the end of the recruitment deadline.
  The surveys inquire into child, parent, and staff perceptions of the waiting space and their overall clinic experience through a mixture of open- and close-ended (e.g. Likert scale) questions.

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Biddiss, PhD, M.A.Sc., Principal Investigator — Holland Bloorview Kids Rehabilitation Hospital; University of Toronto
Locations (1):
- Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario, Canada